CLINICAL TRIAL: NCT02708342
Title: Observational, Retrospective Analysis to Evaluate Switching to Raltegravir Plus Abacavir/Lamivudine in HIV-1-Infected Patients. ORASWIRAL Study
Brief Title: Observational, Retrospective Analysis in HIV-1 Infected Patients. (ORASWIRAL)
Status: Completed | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Castagna Antonella, Professor - (PI and Promoter Professor Adriano Lazzarin), Ospedale San Raffaele
Other Study IDs: ORASWIRAL
Record Dates: First submitted 2016-03-02; First posted 2016-03-15 (Estimated); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: HIV

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
RESEARCH METHODS Study Design Observational, Retrospective, Single-center, Single-arm Study of patients treated with raltegravir plus abacavir and lamivudine.

DETAILED DESCRIPTION:
Adult, male and female HIV-1 infected subjects, who started an antiretroviral regimen of RALTEGRAVIR plus ABACAVIR and LAMIVUDINE after a different antiretroviral regimen.

Subject Selection: Inclusion Criteria

All consecutive patients fulfilling the following inclusion criteria will be considered:

* HIV-1 infected patients,
* age > 18 years,
* Human leukocyte antigen (HLA) B5701-negative
* treatment-experienced patients with viral suppression (HIV-RNA <50 copies/mL), who switched from any antiretroviral drug to raltegravir plus abacavir and lamivudine because of toxicity, convenience or other reasons
* switch from Protease Inhibitor to Raltegravir in patients on Abacavir and lamivudine, switch from any Nucleoside analog reverse-transcriptase inhibitors (NRTI) combination to abacavir and lamivudine in patients on raltegravir, switch to raltegravir plus abacavir and lamivudine from any other combination will all allow the inclusion in the study
* At least one viral load assessed before and at least once after starting the study regimen.

Subject Selection: Exclusion Criteria

* Documented drug-resistance or virological failure to integrase inhibitors, abacavir or lamivudine before starting the study regimen.
* Pregnancy at the start of the study regimen.
* HBsAg positive.

Definitions

Treatment Failure will be defined as the occurrence of Virological Failure or change in any component of the study regimen for any reason or treatment discontinuation at any time after the start of the considered treatment.

Virological failure will be defined by the occurrence of two consecutive (confirmed ) viral loads >50 copies/mL at any time during follow-up.

Variables/Information

The following information will be extracted from the Hospital database of the Department:

* demographics (age, sex, race)
* smoking
* risk factors for HIV infection
* time from HIV-1 diagnosis (years)
* history of AIDS diagnosis
* hepatitis C virus (HCV) co-infection
* hepatitis B virus (HBV) co-infection
* presence of co-morbidities (including diabetes, hypertension, Cardio Vascular Diseases, Chronic kidney disease, cancer, etc)
* reasons for switching to raltegravir + abacavir/lamivudine
* time with HIV-1 RNA < 50 copies/mL before switch
* BMI
* Hematology (Hb, PLT)
* Creatinine
* eGFR epidermal growth factor receptor (Chronic kidney disease -EPI formula)
* Phosphorus
* Calcium
* Aspartate aminotransferase (AST)
* ALT
* FIB-4 (liver index)
* alkaline phosphatase
* total, direct, indirect bilirubin
* proteinuria
* hemoglobinuria
* total, HDL-, LDL-cholesterol
* triglycerides
* glycemia
* HIV-RNA
* lymphocytes (CD4+, CD8+, CD4/CD8 ratio) since the start of raltegravir
* previous antiretroviral regimen and number of previous antiretroviral agents.

Data Sources

The data source is the Infectious Diseases Database of San Raffaele Hospital (IDD-OSR), collecting all the data of patients followed in the outpatient clinic.

Data are collected during routine clinical activity. Adverse Events that occurred after the initiation of the study treatment will be recorded and classified as drug-related or not and according to severity.

Power/Sample Size:

100 patients fulfilling the specified inclusion criteria will be available for this analysis.

When the estimated treatment efficacy proportion is 80%, a sample size of 100 subjects produces a two-sided 95% confidence interval with a precision equal to 8%.

Data Analysis Baseline characteristics of enrolled patients will be described by median and interquartile range or frequency (%), according to the variable type.

Follow-up will count from the date of starting with Raltegravir plus Abacavir and lamivudine to Treatment Failure or last available visit, whichever will first occur.

Primary analysis Kaplan-Meier curves and proportional hazards regression models will be used in reference to the primary endpoint.

Secondary analyses Trend over time of continuous variables (height, weight, BMI, Hb, PLT, creatinine, eGFR, phosphorus, calcium, AST, ALT, FIB-4, alkaline phosphatase, total, direct, indirect bilirubin, total, HDL-, LDL-cholesterol, triglycerides, glycaemia, HIV-RNA, CD4+ cell count) will be assessed by the ANOVA for repeated measures or univariate mixed linear models (depending on the data structure); chi-square test for trend will be applied on categorical variables (proteinuria, hemoglobinuria).

The non-parametric Wilcoxon signed rank test will be applied to assess significant changes of continuous variables since baseline and the last available visit; to test for changes in proportions between baseline and the last available visit, the McNemar test will be calculated.

Relationships among continuous variables (height ,weight, BMI, Hb, PLT, creatinine, eGFR, phosphorus, calcium, AST, ALT, FIB-4, alkaline phosphatase, total, direct, indirect bilirubin, total, HDL-, LDL-cholesterol, triglycerides, glycaemia, HIV-RNA, CD4+ cell count) will be tested calculating the correlation coefficients (Spearman rho, as appropriate).

Safety data analysis will be descriptive only. Adverse Events, Serious Adverse Events will be tabulated, also according to their severity, for a descriptive purpose only.

A two-sided alpha level of 0.05 will be taken as reference to detect statistical significance.

All analyses will be performed with Statistical Analysis Software, release 9.2.

ELIGIBILITY:
Subject Selection: Inclusion Criteria

All consecutive patients fulfilling the following inclusion criteria will be considered:

* HIV-1 infected patients,
* age > 18 years,
* Human leukocyte antigen (HLA) B5701-negative
* treatment-experienced patients with viral suppression (HIV-RNA <50 copies/mL), who switched from any antiretroviral drug to raltegravir plus abacavir and lamivudine because of toxicity, convenience or other reasons
* switch from Protease Inhibitor to Raltegravir in patients on Abacavir and lamivudine, switch from any Nucleoside analog reverse-transcriptase inhibitors (NRTI) combination to abacavir and lamivudine in patients on raltegravir, switch to raltegravir plus abacavir and lamivudine from any other combination will all allow the inclusion in the study
* At least one viral load assessed before and at least once after starting the study regimen.

Subject Selection: Exclusion Criteria

* Documented drug-resistance or virological failure to integrase inhibitors, abacavir or lamivudine before starting the study regimen.
* Pregnancy at the start of the study regimen.
* HBsAg positive.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patient HIV-1 positive treated with raltegravir plus abacavir and lamivudine
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2016-04; Primary Completion 2016-11 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Durability of an antiretroviral regimen of raltegravir plus abacavir and lamivudine | time to treatment failure through 96 weeks

SECONDARY OUTCOMES:
Cumulative probability of virological failure | through 96 weeks
  Kaplan-Meier curves
Proportion of patients with virological failure | through 96 weeks
Proportion of patients with treatment failure | through 96 weeks
Proportion of patients with more or equal to grade 2 abnormal laboratory tests | through 96 weeks
Change in Lymphocytes CD4+ | through 96 weeks
  cells/uL
Change in Lymphocytes CD8+ | through 96 weeks
  cells/uL
Change in Lymphocytes CD4+/CD8+ ratio | through 96 weeks
Changes in total cholesterol | through 96 weeks
  mg/dL
Changes in HDL cholesterol | through 96 weeks
  mg/dL
Changes in LDL cholesterol | through 96 weeks
  mg/dL
Changes in triglycerides | through 96 weeks
  mg/dL
Changes in glucose | through 96 weeks
  mg/dL
Changes in creatinine | through 96 weeks
  mg/dL
Changes in phosphate | through 96 weeks
  mmol/L
Changes in AST | through 96 weeks
  U/L
Changes in ALT | through 96 weeks
  U/L
Changes in ALP | through 96 weeks
  U/L
Changes in FIB-4 (liver index) | through 96 weeks
Changes in eGFR | through 96 weeks
  ml/min/1.73m^2
Changes in proteinuria | through 96 weeks
  mg/dL
Occurrence of HIV genotypic mutations in plasma samples from patients with virological failure | through 96 weeks
Proportion of patients with Adverse events and/or Serious Adverse Events, also according to their severity | through 96 weeks

IPD SHARING:
Plan to Share IPD: Yes
Abstract to Scientific Congress

REFERENCES:
- [Result] Raffi F, Jaeger H, Quiros-Roldan E, Albrecht H, Belonosova E, Gatell JM, Baril JG, Domingo P, Brennan C, Almond S, Min S; extended SPRING-2 Study Group. Once-daily dolutegravir versus twice-daily raltegravir in antiretroviral-naive adults with HIV-1 infection (SPRING-2 study): 96 week results from a randomised, double-blind, non-inferiority trial. Lancet Infect Dis. 2013 Nov;13(11):927-35. doi: 10.1016/S1473-3099(13)70257-3. Epub 2013 Sep 25. PMID 24074642
- [Result] Suzuki A, Uehara Y, Saita M, Inui A, Isonuma H, Naito T. Raltegravir and Abacavir/Lamivudine in Japanese Treatment-Naive and Treatment-Experienced Patients with HIV Infection: a 48-Week Retrospective Pilot Analysis. Jpn J Infect Dis. 2016;69(1):33-8. doi: 10.7883/yoken.JJID.2014.236. Epub 2015 May 12. PMID 25971320
- [Result] Fabbiani M, Mondi A, Colafigli M, D'Ettorre G, Paoletti F, D'Avino A, Ciccarelli N, Sidella L, Murri R, Fortuna S, Vullo V, Cauda R, De Luca A, Di Giambenedetto S. Safety and efficacy of treatment switch to raltegravir plus tenofovir/emtricitabine or abacavir/lamivudine in patients with optimal virological control: 48-week results from a randomized pilot study (Raltegravir Switch for Toxicity or Adverse Events, RASTA Study). Scand J Infect Dis. 2014 Jan;46(1):34-45. doi: 10.3109/00365548.2013.840920. Epub 2013 Oct 28. PMID 24161018
- [Result] Martinez E, d'Albuquerque PM, Perez I, Pich J, Gatell JM. Abacavir/lamivudine versus tenofovir/emtricitabine in virologically suppressed patients switching from ritonavir-boosted protease inhibitors to raltegravir. AIDS Res Hum Retroviruses. 2013 Feb;29(2):235-41. doi: 10.1089/AID.2012.0150. Epub 2012 Sep 24. PMID 22916715
- [Result] Young B, Vanig T, Dejesus E, Hawkins T, St Clair M, Yau L, Ha B, Shield Study Team. A pilot study of abacavir/lamivudine and raltegravir in antiretroviral-naive HIV-1-infected patients: 48-week results of the SHIELD trial. HIV Clin Trials. 2010 Sep-Oct;11(5):260-9. doi: 10.1310/hct1105-260. PMID 21126956
- See also: Italian Guidelines for the management of antiretroviral therapy of the subjects with HIV-1 infection. — http://www.salute.gov.it/portale/temi/p2_6.jsp?lingua=italiano&id=187&area=aids&menu=vuoto